CLINICAL TRIAL: NCT02026154
Title: Finding Early Predictors of Myocardial Dysfunction in Patients With Hypertension - Pilot Study.
Brief Title: Finding Early Predictors of Myocardial Dysfunction
Status: Completed | Type: Observational
Sponsor: Medical University of Lodz (Other)
Responsible Party: Principal Investigator, Agata Bielecka-Dabrowa, MD, PhD, Department of Hypertension, MD, PhD, FESC, cardiologist, Medical University of Lodz
Other Study IDs: RNN/749/13/KB; grant for young scientist 2012 (Other Grant/Funding Number: Polish Cardiac Society)
Record Dates: First submitted 2013-12-31; First posted 2014-01-01 (Estimated); Last update posted 2014-05-06 (Estimated); Status verified 2014-05

CONDITIONS: Hypertension; Heart Failure
Keywords: hypertension, biomarkers, echocardiography, heart failure
MeSH Terms: conditions — Hypertension; Heart Failure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — blood plasma
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- A, B, C: Group A- 15 patients without symptoms of heart failure - control group Group B- 30 patients with exertional dyspnoea Group C - 40 patients with overt heart failure

SUMMARY:
The study objective is to clarify the grounds of heart exertional dyspnoea stenocardia in patients with well-controlled stage I or II hypertension according to European Society of Hypertension, without changes in epicardial coronary arteries in CT coronary angiography and normal resting echocardiography result, and to assess of potential early markers of heart hypertrophy and failure in patients with hypertension.

DETAILED DESCRIPTION:
The study is to allow for identification of patients with hypertension, in whom an early introduction of pharmacological treatment of heart failure HF should be considered. Evaluation in the detection of asymptomatic myocardial dysfunction will include potential heart failure markers such as: cardiotrophin 1, cystatin C, serum syndecan-4, collagen III N-terminal propeptide [PIIINP], NT-proBNP, IL1RL1 and modern echocardiography methods in order to increase the effectiveness of prevention, diagnosis and treatment optimalization.

Material and study plan about 100 persons (age 30-70 years old) will be included in the study, patients with stage I or II primary hypertension according to the European Society of Hypertension: Group A- 15 patients without symptoms of heart failure Group B- 30 patients with exertional dyspnoea Group C - 40 patients with overt heart failure

In group B (patients with exertional dyspnea/stenocardia) we will include only patients who have undergone CT coronary angiography without any identified changes in the epicardial coronary arteries, which will facilitate answering the presented purpose of research. Patients in groups A and B with normal resting echocardiography and treated with a maximum of 2 antihypertensive drugs (an ACE inhibitor or a sartan as therapy base), according to the following regimen:

ACEI/ARB + diuretic ACEI/ARB + calcium channel antagonist Group C - treatment in accordance with the standards for heart failure. Each patient will be informed about the objectives of the study and give written consent to participate.

After signing informed consent patients will have performed the following tests:

* Interview and documentation analysis,
* Physical examination,
* Electrocardiogram
* Echocardiography at rest and during submaximal exercise on a bicycle ergometer
* Levels of markers: cystatin C, cardiotrophin-1, Procollagen III N-Terminal Propeptide (PIIINP), Syndecan 4 (SDC4) and NT-proBNP, IL1RL1. Each patient will be informed about the objectives of the study and give written consent to participate.

ELIGIBILITY:
Inclusion Criteria:

* persons (age 30-70 years old) will be included in the study, patients with stage I or II primary hypertension according to the European Society of Hypertension

Exclusion Criteria:

* with coronary artery disease or a history of coronary artery disease (A, B)
* with unstable hypertension
* with a positive stress test
* with NYHA class III-IV heart failure
* after percutaneous or surgical revascularization
* with diabetes
* with GFR < 60
* with hyperthyroidism and hypothyroidism
* active smokers
* with an implanted pacemaker
* with obesity level II and III
* with ECG-arrhythmia
* pregnant and lactating
* with congenital heart disease
* with hemodynamically significant acquired heart defects
* with cardiomyopathies (A,B)
* with cancer
* with anemia
* abusing alcohol or drugs
* with chronic inflammatory and other diseases
* or who have not given their informed consent to participate in the study

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: persons (age 30-70 years old) will be included in the study, patients with stage I or II primary hypertension according to the European Society of Hypertension
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2012-10; Primary Completion 2014-02 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Number of patients with changes in echocardiography during exercise | 1 year
  Echocardiography at rest and during submaxinal exercise on a bicycle ergometer

SECONDARY OUTCOMES:
Changes in biomarkers levels according to clinical symptoms and echocardiography results | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Agata Bielecka-Dabrowa, PhD, Principal Investigator — Medical University of Lodz
Locations (1):
- Department of Hypertension, Medical University of Lodz, Lodz, Poland